CLINICAL TRIAL: NCT06197646
Title: The Effect of Using Masks With Cartoon Heroes on Treatment Compliance and Parental Satisfaction in Inhaler Therapy Applications in Children
Brief Title: Inhalation Therapy and Therapeutic Play
Acronym: INHALATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23/185
Record Dates: First submitted 2023-12-11; First posted 2024-01-09 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2023-12

CONDITIONS: Inhalation; Respiratory Disease
Keywords: inhaler therapy; children; inhalation; therapeutic play; nursing
MeSH Terms: conditions — Respiratory Aspiration; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaler mask with cartoon characters (Experimental): Inhalation therapy with cartoon characters inhaler mask and Inhaler therapy training
  Interventions: Device: Cartoon characters inhaler mask
- Inhaler mask (No Intervention): Inhalation therapy with the inhaler mask routinely used by the clinic and Inhaler therapy training

INTERVENTIONS:
Device: Cartoon characters inhaler mask — Cartoon characters inhaler mask
  Arms: Inhaler mask with cartoon characters

SUMMARY:
The aim of this clinical research study was to determine the effect of the use of a cartoon character mask on treatment compliance and parental satisfaction and to evaluate the effectiveness of the cartoon character mask in children receiving inhaled therapy for the treatment of respiratory system diseases in children.

The hypotheses it aims to answer are as follows:

H1: Inhalers given using a mask with a cartoon character facilitate treatment compliance.

H2: The inhaler given using a mask with a cartoon character makes treatment compliance difficult.

H3: Inhaler treatment using a mask with a cartoon hero increases parental satisfaction.

H4: Inhaler treatment using a mask with a cartoon hero decreases parental satisfaction.

H5: Inhaler treatment using a mask with a cartoon hero has a positive effect on the hospitalization process.

H6: Inhaler treatment using a mask with a cartoon hero has a positive effect on the recovery process.

H7: Compared to routine inhaler mask use, the use of masks with cartoon heroes provides a positive relationship between treatment adherence and parental satisfaction.

In the study, according to randomization, the intervention group will receive inhalers with masks, and the other group will receive inhalers routinely used in the clinic. The treatment of the children was planned by the physician, and no additional treatment was given for the study. Children's adherence to treatment and parents; satisfaction will be evaluated. The effectiveness of the masked inhaler used will be asked.

DETAILED DESCRIPTION:
Respiratory diseases are among the most common diseases in childhood and are among the most important causes of infectious disease-related mortality and morbidity worldwide. Approximately 1 in 3 children have a lower respiratory tract infection in the first year of life. Respiratory tract infections are more common in developing countries and have a worse prognosis. According to World Health Organization data, respiratory tract infections constitute 13% of the causes of mortality in children under 5 years of age. Respiratory tract diseases are frequently seen during seasonal transitions in childhood and are caused by viral or bacterial agents. Treatment of respiratory tract diseases differs as outpatient or inpatient depending on the agent and the condition of the child. In addition to antibiotherapy, relaxing and supportive treatments are also included in the treatment. These include analgesics, antipyretics, decongestants, and antihistamines. These treatments are administered orally, parenterally, or inhaled. In inhaler treatment, medication is given by placing it into a pediatric mask with a reservoir. This treatment method is boring, frightening, and anxiety-inducing for the pediatric age group and makes it difficult to comply with the treatment. Various methods are being tried to facilitate compliance with treatment in children. One of these methods is play-based treatment activities.

Play is a form of learning that facilitates children's adaptation to the outside world by providing them with new experiences, skills, and social responsibility, and enables them to communicate by exploring their environment. Play is defined by the United Nations High Commission for Human Rights as the right of every child that contributes to the development of the child. In the literature, it is reported that play is effective in reducing the anxiety and fear of hospitalized children and is necessary to provide holistic and quality care. It has also been reported that it does not benefit their recovery by relaxing them both physically and emotionally.

Games are categorized under four headings according to their purpose: entertaining and distracting games, games that support the development of cognitive, social, and sensorimotor skills, games that teach right and wrong, provide socialization, make people aware of and accept their biological existence as men or women, and therapeutic games to relieve anxiety and tension. Games can be used in clinics as healing practices (therapeutic practices). Although therapeutic play and play therapy are used interchangeably, they are conceptually and practically quite different. The spontaneous creation of activities using toys without predetermined goals is referred to as play therapy.

Therapeutic play that activates physiological functions is used in cases where the child exhibits regressive behavior, drama therapeutic play that allows emotional discharge, and educational/creative therapeutic play is used to prepare children for procedures.

There are three types of therapeutic play:

1. Energy Expending Play: Children show their aggressive behavior, anger, and anxiety by shouting, punching, and running. To direct these emotions in the hospital, areas for this purpose should be created or appropriate materials should be provided. In this way, their aggressive behavior, anger, and anxiety levels can be reduced.
2. Dramatic Play: Playing by imitating life and events to understand them better is defined as dramatic play.

   By using dramatic play, it is ensured that the child expresses his/her feelings about the interventions to be applied in the hospital environment and major events. For this purpose, playing with medical equipment such as masks, stethoscopes, and IV sets during the game can be effective in reducing the stress of children and expressing what they feel.
3. Creative Play: This is the type of play used to show children how each procedure is done by using materials before and after the procedures. In creative play, methods such as drawing pictures, sentence completion, and three wishes tests are used to collect information about the inner world of the child.

The main aim of the therapeutic relationship in pediatric nursing is to maintain the health, growth, and development of the child and his/her family at the highest possible level. Nurses help children and their parents to maintain their health and develop adaptation by gaining effective coping skills in case of illness or any lifestyle change.

Nurses can use play as a health care strategy for hospitalized children in three areas. The first of these areas is its use in routine practices. Secondly, it is recommended to use it in preparation for surgical or invasive interventions and finally during painful and unpleasant procedures.

For nurses, play is key to understanding the child. Therapeutic play helps children to express their feelings and thoughts verbally or non-verbally about the procedures to be applied. The nurse adapts therapeutic play to care and provides nursing care in line with the information gathered through play. Florence Nightingale, the founder of modern nursing, emphasized the necessity of play for hospitalized children. Studies have reported that therapeutic play practice contributes to holistic and specific nursing care and that therapeutic play is an effective method. However, it was found that most of them did not use it in daily nursing practices due to reasons such as lack of time.

In the last decade, it has been known that showing videos and distributing booklets and coloring books to children at the pre-anesthetic visit is beneficial. Arranging the anesthesia mask to resemble popular characters among children (such as birds, and cartoon characters), having children put the masks on their faces and look at the fun face mask in the mirror and blowing on the balloon, making it look like a magic ball, allowing children to stick the stickers they like on the anesthesia mask as a game facilitates induction of anesthesia. With pharmacological premedication appropriate to these nonpharmacological methods, anxiety can be prevented, psychological injuries can be reduced, induction of anesthesia can be facilitated, and preoperative anxiety of the child can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 3-12
* Being in a pediatric clinic
* Being diagnosed with respiratory system diseases
* Being on inhaler therapy as part of routine treatment
* Self and parent's consent to participate in the study

Exclusion Criteria:

* Having a cognitive or neurological problem
* Not taking inhaler therapy routinely
* Being a foreign national

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Treatment compliance | 6 months
  The primary outcome of the study will be to determine children's compliance with inhalation therapy with an inhaler mask.

SECONDARY OUTCOMES:
Effectiveness and usefulness of the treatment tool | 6 months
  As a secondary result, the effectiveness and usefulness of the cartoon character mask developed within the framework of therapeutic play will be evaluated.

OTHER OUTCOMES:
Parental satisfaction | 6 moths
  As a tertiary outcome, parental satisfaction with the applied method will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Simsek, Study Director — Istinye University
Locations (1):
- Istinye University, Istanbul, Zeytınburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Once completed, the study will be published in a scientific journal. After publication, IPD will be shared upon request.
  Researchers will have access to the IPD. The materials and methods section will be shared upon reasonable request.

REFERENCES:
- [Background] undefined
- [Background] Gül, O. (2015). The effect of game on pre-school period (ages 3-6): A review of study. Turkish Journal of Sport and Exercise, 17(3), 1. https://doi.org/10.15314/tjse.
- [Background] Ginsburg KR; American Academy of Pediatrics Committee on Communications; American Academy of Pediatrics Committee on Psychosocial Aspects of Child and Family Health. The importance of play in promoting healthy child development and maintaining strong parent-child bonds. Pediatrics. 2007 Jan;119(1):182-91. doi: 10.1542/peds.2006-2697. PMID 17200287
- [Background] Francischinelli, A. G., Almeida, F. A. &, & Fernandes, M. S. (2012). Routine use of therapeutic play in the care of hospitalized children: nurses' perceptions. Acta Paul Enferm, 25(1), 18-23. https://doi.org/10.1590/S0103- 21002012000100004
- [Background] Çavuşoğlu H. (2013). Child Health Nursing. Ankara: System Ofset Printing House: p. 67-69
- [Background] Çiftçi, E. N. (2011). The effect of visual and auditory premedication on mask induction in children. Trakya University, Faculty of Medicine, Specialization Thesis (Advisor Sevtap Hekimoğlu Şahin), Edirne.
- [Background] Berna, I. K., Ceren, Ç., & Esenay Figen. (2013). Therapeutic play: the key to communication with the sick child. Ankara Journal of Health Sciences, 2(123), 1-10. https://doi.org/10.1501/Asbd_0000000038
- [Background] Aydın T, Şahin L, Algın C, Kabay Ş, Yücel M, Hacıoğlu A et al. Do not mask the mask: use it a premedicant. Pediatric Anesthesia 2008;18:107-12.
- [Background] Altay, N. C. (2008). Preoperative preparation in children. Hacettepe University Faculty of Health Sciences Nursing Journal, 68-76.
- [Result] Koukourikos K, Tzeha L, Pantelidou P, Tsaloglidou A. THE IMPORTANCE OF PLAY DURING HOSPITALIZATION OF CHILDREN. Mater Sociomed. 2015 Dec;27(6):438-41. doi: 10.5455/msm.2015.27.438-441. PMID 26889107